CLINICAL TRIAL: NCT03168984
Title: A Single-Centre, Investigator/Subject Blind, Placebo-Controlled, Single and Multiple Oral Dose Investigation of Safety, Tolerability, and Pharmacokinetics of UCB0942 in Healthy Japanese and Caucasian Subjects
Brief Title: A Study to Investigate the Safety, Tolerability, and Pharmacokinetics of UCB0942 in Healthy Japanese and Caucasian Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: UP0039; 2017-000385-30 (EudraCT Number)
Record Dates: First submitted 2017-05-17; First posted 2017-05-30 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Healthy Japanese and Caucasian Subjects
Keywords: Healthy Japanese subjects; Healthy Caucasian subjects; UCB0942

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UCB0942 (Experimental): Cohort 1 (Japanese subjects): Single dose of UCB0942 (dosage regimen 1) Cohort 2 (Japanese subjects): Single dose of UCB0942 (dosage regimen 2) Cohort 3 (Japanese subjects): Single dose of UCB0942 (dosage regimen 3) followed, after maximum 21 days, by multiple doses of UCB0942 (dosage regimen 2) Cohort 4 (Caucasian subjects): Single dose of UCB0942 (dosage regimen 3) followed, after maximum 21 days, by multiple doses of UCB0942 (dosage regimen 2)
  Interventions: Drug: UCB0942
- Placebo (Placebo Comparator): Cohort 1 and Cohort 2: Single dose of Placebo Cohort 3 and Cohort 4: Single dose of Placebo followed, after maximum 21 days, by multiple doses of Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: UCB0942 — * Pharmaceutical form: Film-coated tablet
  * Route of administration: Oral use
  Arms: UCB0942
Other: Placebo — * Pharmaceutical form: Film-coated tablet
  * Route of administration: Oral use
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the pharmacokinetics, safety and tolerability of UCB0942 in Japanese and Caucasian subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female and between 20 and 55 years of age (inclusive)
* Subject is in good physical and mental health
* Female subjects will use an efficient form of contraception for the duration of the study (unless menopausal)
* Male subject agrees that, during the study period, when having sexual intercourse with a woman of childbearing potential, he will use an efficient barrier contraceptive AND that the respective partner will use an additional efficient contraceptive method
* For Japanese subjects: Subject is of Japanese descent as evidenced by appearance and verbal confirmation of familial heritage (a subject has all 4 Japanese grandparents born in Japan)
* For Caucasians: Subject is of Caucasian descent as evidenced by appearance and verbal confirmation of familial heritage (a subject has 4 Caucasian grandparents).

Exclusion Criteria:

At screening:

* Previous study participation with another investigational medicinal product (IMP) within 3 months
* History of alcohol/drug abuse
* History of psychiatric condition and suicide attempt
* Any medical condition unfit for study (including history of cancer)
* History of hypersensitivity for IMP components
* Taking concomitant medications
* Positive for human immunodeficiency virus (HIV)/ hepatitis B virus (HBV)/ hepatitis C virus (HCV)
* Abnormal liver function tests (LFTs), abnormal safety bloods/ vitals/ physical examination and electrocardiogram (ECG) findings
* Positive for pregnancy test
* Other protocol-defined exclusion criteria may apply

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2017-08-14 (Actual); Study Completion 2017-08-14 (Actual)

PRIMARY OUTCOMES:
Cmax: maximum observed plasma concentration of UCB0942 and metabolites | Plasma will be collected predose and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, and 48 hours postdose.
AUC(0-t): area under the plasma concentration-time curve from time zero to the time of last detectable concentration for UCB0942 and metabolites | Plasma will be collected predose and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, and 48 hours postdose.

SECONDARY OUTCOMES:
tmax: time of maximum concentration of UCB0942 and metabolites during the Single-dose period | Plasma will be collected predose and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, and 48 hours postdose.
tmax: time of maximum concentration of UCB0942 and metabolites during the Multiple-dose period | Plasma will be collected predose and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, and 48 hours postdose.
AUC: area under the plasma concentration-time curve from time zero to infinity for UCB0942 and metabolites during the Single-dose period | Plasma will be collected predose and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, and 48 hours postdose.
  AUC is calculated as AUC(0-t)+Clast/kel, where Clast is the last observed quantifiable plasma concentration and kel is the apparent terminal elimination rate constant
t1/2: apparent terminal elimination half-life of UCB0942 and metabolites during the Single-dose period | Plasma will be collected predose and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, and 48 hours postdose.
t1/2: apparent terminal elimination half-life of UCB0942 and metabolites during the Multiple-dose period | Plasma will be collected predose and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, and 48 hours postdose.
RCmax: Accumulation ratio of Cmax for UCB0942 and metabolites during the Multiple-dose period | Plasma will be collected predose and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, and 48 hours postdose.
AUCtau: area under the curve over a dosing interval (12hrs) for UCB0942 and metabolites during the Single-dose period | Plasma will be collected predose and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, and 48 hours postdose.
AUCtau: area under the curve over a dosing interval (12hrs) for UCB0942 and metabolites during the Multiple-dose period | Plasma will be collected predose and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, and 48 hours postdose.
RAUC: Accumulation ratio of AUCtau for UCB0942 and metabolites during the Multiple-dose period | Plasma will be collected predose and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, and 48 hours postdose.
Adverse events (AEs) reported spontaneously by the subject or observed by the investigator | From Screening until safety follow up visit (up to Week 18)
Change from baseline in laboratory variables, vital sign variables, 12-lead ECG variables and physical examination | From Baseline until safety follow up visit (up to Week 18)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 844 599 2273 (UCB)
Locations (1):
- Up0039 001, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No